CLINICAL TRIAL: NCT02441335
Title: CellulaR Injury and Preterm Birth
Acronym: CRIB
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: March of Dimes (Other)
Responsible Party: Sponsor
Other Study IDs: 821376
Record Dates: First submitted 2015-04-06; First posted 2015-05-12 (Estimated); Last update posted 2019-10-07 (Actual); Status verified 2019-10

CONDITIONS: Preterm Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. Collect blood, urine and cervicovaginal cells from women with preterm labor and term labor in order to investigate:
  1. What is the role of bioenergetics in pregnancy and what are the pertubations in cell metabolism that lead to spontaneous preterm birth
  2. What are the interactions between the microbiome (oral, gut, cervicovaginal, and placental) and host metabolic function in pregnancy
  3. How do interactions between cell metabolism and the microbiome influence cervical remodeling and placental function leading to spontaneous preterm delivery
  4. What genetic and environmental factors influence the metabolic function of reproductive tissues leading to spontaneous preterm delivery
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group 1 (Preterm labor, PPROM, cervical insufficiency): Singleton pregnancy between 20 0/7 36 6/7 weeks gestational age who is admitted with PTL or cervical insufficiency (Equal or greater than 2 cm dilated) or PPROM
- Group 2 (Term labor): Admitted to the hospital with spontaneous labor (regular contractions, cervical dilation) or spontaneous rupture of membranes
- Group 3 (PTB-medically indicated): Singleton pregnancy between 20 0/7 34 5/6 weeks gestational age who is admitted with a medically indicated preterm birth (IOL for abruption, non reassuring fetal heart tones, intrauterine growth restriction, preeclampsia, trauma, etc.)

SUMMARY:
The goal of this study is to examine how cellular dysfunction can lead to preterm birth. Women with singleton pregnancies with spontaneous preterm labor, preterm premature rupture of membranes, and cervical insufficiency (20 to 36-6/7 weeks gestation), and term deliveries (greater than 38 weeks) will be enrolled. Medical/obstetric history and pregnancy outcomes will be recorded. Maternal blood, urine and cervical cells (enrollment); cord blood and placental biopsy (delivery) will be collected.

DETAILED DESCRIPTION:
Despite improvements in prenatal care, preterm birth (PTB) remains a leading contributor to perinatal morbidity and mortality. Several genetic and environmental factors have been associated with spontaneous preterm birth, but the pathways by which these factors induce preterm delivery have not been defined. The March of Dimes CPR at the University of Pennsylvania was created to help elucidate the pathogenesis of preterm birth by bringing together a diverse team of investigators with expertise in preterm birth, cellular metabolism, genetics, mitochondrial functional analyses, genome, epigenome, and transcriptome profiling, integrated bioinformatics analyses, and microbiome research. The center will focus on addressing the interactions between bioenergetics, genetics, microbiome, abnormal cervical remodeling and placental dysfunction. Each one of these factors will be studied independently and in relation to the other factors. In order to study metabolic processes in relation to spontaneous PTB, a prospective case-control study will be performed. This study will involve women with singleton pregnancies with spontaneous preterm labor (PTL), preterm premature rupture of membranes (PPROM), and cervical insufficiency, between 20-0/7 and 36-6/7 weeks gestational age (cases), and women with term deliveries (38 to 41 weeks gestation, controls). The investigators will obtain information regarding the patients' pertinent past medical and obstetric histories, and the following specimens will be collected: maternal blood, maternal urine, and cervical epithelial cells at enrollment; and umbilical cord blood and placental biopsies at delivery. We will follow and record each of these patients' pregnancy outcomes.

ELIGIBILITY:
Cases:

Inclusion Criteria:

* 18-45 years of age
* Singleton pregnancy between 20 0/7 and 36 6/7 weeks gestational age who is admitted with preterm labor or cervical insufficiency (greater than 2 cm dilation) or Preterm Premature Rupture of Membranes

Exclusion Criteria:

* Multiple gestation
* Fetal chromosomal abnormality
* Major fetal anomaly
* Intra-uterine fetal demise
* Gestational hypertension/preeclampsia

Controls:

Inclusion Criteria:

* 18-45 years of age
* Singleton pregnancy that delivers at term (38 to 41 weeks gestational age)
* Admitted to the hospital with spontaneous labor (regular contractions, cervical dilation) or spontaneous rupture of membranes

Exclusion Criteria:

* Multiple gestation
* Fetal chromosomal abnormality
* Major fetal anomaly
* Intra-uterine fetal demise
* Intra-uterine growth restriction
* Gestational hypertension/preeclampsia
* Clinical chorioaminionitis
* Induction of labor
* Elective c-section

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: At HUP, there are approximately 4,200 deliveries a year, of which approximately 10 percent (420) deliver preterm. Among these preterm births, two-thirds (280) are spontaneous, which is the focus of our research. Many women who ultimately have a preterm birth, first present with preterm labor. Women who have advanced dilatation, preterm rupture of membranes, etc are at high risk for having a preterm birth. The investigators anticipate, based on the number of spontaneous preterm births at HUP per year, enrolling about 40-50% of those eligible and understanding that about 40% of those enrolled will have a preterm birth, we should be able to enroll about 112 women per year over 5 years. The coordinators will enroll cases who are admitted to the hospital with PTL, PPROM, or cervical insufficiency at 20-0/7 to 36-6/7 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 705 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Biogenetics | 5 years
  The role of biogenetics in pregnancy and what are the perturbations in cell metabolism that lead to spontaneous preterm birth.
Microbiome | 5 years
  The interactions between the microbiome (oral, gut, cervicovaginal, and placental) and host metabolic function in pregnancy.
Cervical remodeling | 5 years
  How the interactions between cell metabolism and the microbiome influence cervical remodeling and placental function leading to spontaneous preterm delivery.
Genetics and Environmental factors | 5 years
  How genetic and environmental factors influence the metabolic function of reproductive tissues leading to spontaneous preterm delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Michal Elovitz, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States